CLINICAL TRIAL: NCT01522352
Title: Comparison of Short and Mid-term Hemodynamic Performance Between Three Types of Stented Pericardial Aortic Valves
Brief Title: Comparison Between Three Types of Stented Pericardial Aortic Valves
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Edwards Lifesciences (Industry); Abbott Medical Devices (Industry); Sorin group, Italy (Unknown); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Model: Parallel | Masking: None
Other Study IDs: CHU-0109
Record Dates: First submitted 2011-12-20; First posted 2012-01-31 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Aortic Valve Replacement
Keywords: Bioprosthesis,; aortic valve replacement; Magna Ease; Mitroflow; Trifecta

ARMS (1):
- pericardial aortic valves (Experimental): Comparison of short and mid-term hemodynamic performance between three types of stented pericardial aortic valves: Trifecta aortic valve (St. Jude Medical), Mitroflow aortic valve (Sorin Group), Magna Ease (Edwards Lifesciences)
  Interventions: Procedure: Aortic valve replacement by bioprosthesis

INTERVENTIONS:
Procedure: Aortic valve replacement by bioprosthesis — Comparison of short and mid-term hemodynamic performance between three types of stented pericardial aortic valves: Trifecta aortic valve (St. Jude Medical), Mitroflow aortic valve (Sorin Group), Magna Ease (Edwards Lifesciences)

SUMMARY:
This study suggests for the first time a comparison of the hemodynamic performance of the two most implanted aortic bioprosthesis in France with the new aortic bioprosthesis available since September 2010 at the University Hospital of Clermont Ferrand.

DETAILED DESCRIPTION:
According to the French database Society for Thoracic and Cardiovascular Surgery, 11,621 patients underwent aortic valve replacement in 2007. Over 77% of biologic prosthetic valves were used. Among these biologic valves, those in pericardium are mainly used in all French cardiac surgery centers.

Since March 2010, a new pericardial aortic valve has obtained a CE mark, allowing cardiac surgery centers in Europe to implement it in humans.

Hemodynamic performance of different biologic valves has never been measured. This study suggests for the first time a comparison of the hemodynamic performance of the two most implanted aortic bioprosthesis in France with the new aortic bioprosthesis available since September 2010 at the University Hospital of Clermont Ferrand.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 85 years who need aortic valve replacement (no endocarditis) With Bioprosthesis, with or without myocardial revascularization, with or without tricuspid valve repair surgery

Exclusion Criteria:

* no endocarditis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
measurement of postoperative trans-valvular mean gradient by echocardiography | after 6 months

SECONDARY OUTCOMES:
Comparison between aortic annulus diameter measurement by preoperative CT angiography, transthoracic echocardiography and the aortic annulus' surgical size | at six months
Comparison between the aortic annulus measurement and the implanted bioprosthesis size | at six months
Surgical outcome at hospital | at 6 months.
Postoperative trans-valvular mean gradient by echocardiography | at six months.
Comparison of the transthoracic echocardiography estimated postoperative aortic surfaces | at six months.

CONTACTS AND LOCATIONS:
Overall Officials: Kasra AZARNOUSH, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Azarnoush K, Pereira B, Duale C, Dorigo E, Farhat M, Innorta A, Dauphin N, Geoffroy E, Chabrot P, Camilleri L. Comparison between three types of stented pericardial aortic valves (Trivalve trial): study protocol for a randomized controlled trial. Trials. 2013 Dec 3;14:413. doi: 10.1186/1745-6215-14-413. PMID 24299218